CLINICAL TRIAL: NCT01358162
Title: A Phase 1C, Randomized, Placebo-Controlled, Double-Blinded Study to Evaluate the Safety, Tolerability and Pharmacokinetics of 300 mg of SQ109 Given Once Daily for 14 Days in Normal, Healthy Male and Female Volunteers
Brief Title: Phase IC Study of Safety and PK of SQ109 300mg Daily
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-0111; N01AI80024C
Record Dates: First submitted 2010-11-18; First posted 2011-05-23 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-05

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- SQ109 (Experimental): 300 mg of SQ109, orally, given daily for 14 consecutive days
  Interventions: Drug: SQ109
- Placebo (Placebo Comparator): Placebo given orally, daily for 14 consecutive days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo given orally, daily for 14 consecutive days
  Arms: Placebo
Drug: SQ109 — A single oral dose of 300 mg of SQ109 given daily for 14 consecutive days.
  Arms: SQ109

SUMMARY:
Healthy male and female volunteers will be given SQ109 300mg daily for 14 days to assess the safety and tolerability and pharmacokinetics.

DETAILED DESCRIPTION:
This is a Phase 1C randomized, placebo controlled, double-blinded, in-patient trial of a single oral dose of 300 mg of SQ109 given daily for 14 consecutive days to evaluate the safety, tolerability and pharmacokinetics of SQ109 in normal healthy male and female subjects 18-45 years of age.

Each subject will receive 300 mg of SQ109 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 45 years of age (inclusive).
* Subject must be a healthy male or female volunteer (i.e., hematology, coagulation, clinical chemistries and urinalysis tests must be within study-defined ranges (See Appendix B). Clinical tests must be performed within 28 days of receiving first dose of study drug.
* Body Mass Index (BMI) must be between 18 and 30 kg/m2 inclusive.
* Subject must be Tuberculin Skin Test/Purified Protein Derivative (TST/PPD) negative (within the previous 1 year) at Screening. The TST/PPD may be omitted if the subject presents written evidence of having a negative test during the previous 12 months.
* Subject must be able to give voluntary written informed consent before any study related procedure is performed.
* If female, has no childbearing potential or agrees to avoid becoming pregnant from the day of screening through their entire participation in the trial (Day 28) by using one of the following acceptable methods of birth control plus recommended use of a barrier method (condom) by the male partner (even if vasectomized):

  1. intrauterine contraceptive device; or
  2. diaphragm in combination with contraceptive jelly, cream, or foam; or
  3. spermicide; or
  4. abstinence. Non-childbearing potential is defined as being post-menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy or status after hysterectomy.

Hormonal contraceptives of any type or form (including oral, transdermal, vaginal or depot preparations) will not be allowed during the study.

* All female subjects of childbearing potential must have a negative serum pregnancy test at screening and within 24 hours of the first dose of study product.
* Male subjects must agree to use an acceptable barrier method for birth control (abstinence or use of a condom with spermicide) from screening through Study Day 28 and advice and recommend use of additional birth control (as in criterion 6 above) to female sex partners throughout the study.
* Subject agrees not to donate blood during the study and up to 30 days after Study Day 28.
* Subject agrees to comply with all study requirements, including clinic house rules.

Exclusion Criteria:

* A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Principal Investigator (PI), would jeopardize the safety of the subject or impact the validity of the study results.
* Subject has been on an abnormal diet during the 4 weeks preceding the study. Abnormal diet is defined as a diet in which the subject has a significant change in eating habits (e.g., liquid diet only) and an unbalanced diet (e.g., protein only, high fat, low carbohydrate, etc.).
* Subject has received an investigational drug in a clinical trial within 30 days prior to study initiation.
* Subject has used any OTC medication, including vitamins and herbal supplements, within 7 days prior to Day 1 of the study, unless in the opinion of the PI, the substance would not likely impact on the conduct of this study, including PK of SQ109.
* Subject has used any prescription medication within 14 days prior to Day 1 of the study, or the use of hormonal preparations containing sex hormones within 30 days prior to Day 1 of the study.
* Subject has any current medical condition requiring treatment with medication, either prescription or OTC.

Subject has been treated with any known CYP450 enzyme altering drugs such as azoles, antifungals, barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to Day 1 of the study.

* Subject has a positive blood screen for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody and/or a positive history for alcohol abuse or dependence and/or a positive serum ethanol or a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine metabolites, marijuana, opiates, phencyclidine (PCP)).
* Subject has a baseline QTcF interval >450 msec (males) or >470 msec (females) (defined in Section 9.1.3) or a family history of prolonged QTcF syndrome or premature cardiac death.
* Subject has Wolf Parkinson White Syndrome (WPW) or family history of WPW or a history of supra-ventricular tachycardias or syncope.
* Subject has lived with a person having active TB or has traveled to an area of endemic TB within the past 12 months.
* Subject has an abnormal result on the Ishihara color test, the funduscopic exam, current optic neuritis or known retinal disease.
* Subject has an uncontrolled intercurrent illness (i.e., active infection) or fever (oral temperature >/=100 degrees F or >/= 37.7 degrees C).
* Subject has had major surgery within 4 weeks of study entry.
* Women who are pregnant or breastfeeding.
* Subject has donated blood within the past 30 days prior to Day 1 of the study.
* Subject has allergy to ethambutol or related compounds.
* Subject is an employee of or family member of an employee of Sequella, Quintiles, or DynPort Vaccine Company LLC (DVC).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability via: physical exams, color and visual acuity tests, funduscopic exams, neurological exams, vital signs, electrocardiograms, routine clinical labs (includes chemistry, hematology, coagulation and urinalysis data), and adverse events. | Days 1-14, 16-18, 21 and 28

SECONDARY OUTCOMES:
Pharmacokinetics of SQ109: Serial blood samples prior to and following single/multiple doses: AUC(0-t): area under the concentration time curve to the last time with concentration greater than or equal to the validated limit of quantitation of the assay | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on day 1.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: AUC(0-infinity): area under the concentration time curve to infinity | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on day 1.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: AUC(0-24): area under the concentration time curve to 24 hours | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 1, 5, & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: t1/2: apparent terminal half-life | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 1 & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: CL/F: apparent oral clearance | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 1, 5, & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: Vz/F: apparent volume of distribution | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 1, 5, & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: Cmin: observed minimum concentration | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 5, & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: Cavg: calculated average concentration during the dosing interval | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 5, & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: Tmax: Time of maximum concentration (Cmax) | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 1, 5, & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: AUC(0-tau) Area under the concentration time curve to the end of the dosing interval, 24 hours | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 1, 5, & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: RCmax: Accumulation ratio for Cmax estimated as Cmax (Day 14) / Cmax (Day 1) | Before and after dosing on days 1-14. Serial PK after dosing on days 1 & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: Tmin: Time to minimum concentration (Cmin) | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 1, 5, & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: Linearity Index: AUC(0-tau) (Day 14) / AUC(0-infinity)(Day 1) | Before and after dosing on days 1-14. Serial PK after dosing on days 1 & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: RAUC : Accumulation ratio for AUC estimated as AUC0-tau (Day 14)/ AUC(0-24)(Day 1) | Before and after dosing on days 1-14. Serial PK after dosing on days 1 & 14.
Pharmacokinetics of SQ109: Serial blood samples for measurement of plasma levels of SQ109 prior to and following single/multiple doses: Cmax: observed maximum concentration | Before and after dosing on days 1-14, then on days 16-21 & 28. Serial PK after dosing on days 1, 5, & 14.

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase I Services - Overland Park, Overland Park, Kansas, United States